CLINICAL TRIAL: NCT01190618
Title: Surgical Outcomes of Vaginal Prolapse Repair With the Elevate Prolapse Repair Kit
Brief Title: Surgical Outcomes of Vaginal Prolapse Repair With Elevate
Status: Completed | Type: Observational
Sponsor: Larry Sirls (Other)
Responsible Party: Sponsor-Investigator, Larry Sirls, Principal Investigator, Corewell Health East
Organization: Corewell Health East (Other)
Other Study IDs: 2010-176
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Vaginal Prolapse
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate outcomes in patients having vaginal prolapse repair with the Elevate prolapse repair kit and compare these outcomes to patients who had a repair with Prolift. .

DETAILED DESCRIPTION:
The investigators hypothesize that the less invasive Elevate mesh results in a shorter operative time, lower blood loss, complications, postoperative pain and earlier discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Women who have had a vaginal repair with Elevate prolapse repair kit

Exclusion Criteria:

* N/A

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women having vaginal repair with Elevate prolapse repair kit
Sampling Method: Non-Probability Sample
Enrollment: 417 (Actual)
Dates: Start 2010-08; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of Outcomes | 3 Months
  To evaluate outcomes in patients having vaginal prolapse repair with the Elevate prolapse repair kit and compare these outcomes to patients who had a repair with Profift.

CONTACTS AND LOCATIONS:
Overall Officials: Larry Sirls, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No